CLINICAL TRIAL: NCT00811655
Title: Phase II Single-arm Study of Pre-operative Stereotactic Radiosurgery for Brain Metastases.
Brief Title: Stereotactic Radiosurgery in Treating Patients With Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006870; P30CA014236 (NIH); DUMC-PRO00006870; CDR0000630230 (Other: NCI)
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-10

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: tumors metastatic to brain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pre-Operative SRS (Experimental): SRS pre-operatively with the planned target volume defined as the tumor plus a 3-mm margin.
  Interventions: Procedure: therapeutic conventional surgery; Radiation: stereotactic radiosurgery

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Surgery of a single brain metastasis.
Radiation: stereotactic radiosurgery — Pre-operative single fraction SRS

SUMMARY:
RATIONALE: Stereotactic radiosurgery may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Giving stereotactic radiosurgery before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well stereotactic radiosurgery works in treating patients with brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the rate of recurrence at the surgical site in patients with brain metastases treated with neoadjuvant stereotactic radiosurgery (SRS) compared with historical data documenting recurrence at the surgical site after surgical resection and whole-brain radiotherapy (WBRT).

Secondary

* To estimate the rate of salvage WBRT, SRS, or surgery in patients treated with neoadjuvant SRS alone.
* To determine the volume of adjacent normal brain parenchyma irradiated in these patients.
* To estimate the rate of new brain metastases outside of the neoadjuvant SRS site in these patients.
* To estimate the quality of life of these patients after neoadjuvant SRS alone.
* To assess the effect of SRS and surgical intervention on the preservation of neurocognitive functioning in these patients.
* To determine the clinical significance (mass effect, cognitive functioning, and other symptoms) of locally recurrent brain metastases at the time of their occurrence in these patients.
* To estimate the rate of death due to neurologic causes, defined as death attributable to the progression of neurological disease, in these patients.
* To estimate the overall survival of these patients.

OUTLINE: Patients undergo stereotactic radiosurgery over 30 to 90 minutes. Approximately 2-4 weeks later, patients undergo surgical resection of brain metastasis.

Quality of life and neurocognitive function are assessed periodically using the FACT-Br subscales and Mini-Mental State Exam.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of brain metastases from an extracranial primary site

  * Tumor ≤ 4 cm in maximal extent in any plane on contrast MRI
* Scheduled to undergo gross total resection of a single brain metastasis confirmed by histology

  * Up to 4 metastases allowed provided the largest mass is amenable to surgical resection and all non-resected masses are amenable to stereotactic radiosurgery (SRS)
* RTOG Recursive Partitioning Analysis (RPA) class 1 or 2, as defined by the following:

  * RPA class 1: Karnofsky performance status (KPS) 70-100%; age < 65 years; controlled primary disease; and no extracranial metastatic disease
  * RPA class 2: KPS 70-100%; uncontrolled primary disease; and/or extracranial metastatic disease
* No lesion located in anatomic regions that are not amenable to SRS, including the brain stem, optic apparatus, or eloquent cortex
* No primary lesion with radiosensitive histology (e.g., small cell carcinoma, germ cell tumors, lymphoma, leukemia, or multiple myeloma)
* No radiographic or cytologic evidence of leptomeningeal disease

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* Not pregnant or nursing
* Negative pregnancy test
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Psychiatric illness
* No contraindication to SRS, whole-brain radiotherapy, or MRI

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior brain surgery other than resection of metastasis
* No prior brain radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H. Sampson, MD, PhD, Principal Investigator — Duke University; Hamidreza Aliabadi, MD, Principal Investigator — Duke University; John P. Kirkpatrick, MD, Principal Investigator — Duke University; James E. Herndon, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were consented and interviewed in a private room in the Duke clinics. The patients came to Duke Radiology Center, found to be eligible and then provided options by the neuro-radiologist. They were consented by the research nurse at one of these visits.
Pre-assignment Details: The only reason that enrolled participants were excluded from the trial prior to treatment assignment was if there were development of any exclusion criteria.
Groups:
- Pre-Operative SRS: Stereotactic radiosurgery (SRS) will be administered pre-operatively as a single fraction with the planned target volume defined as the gross tumor volume plus a 3mm margin.
  therapeutic conventional surgery : Surgery of a single brain metastasis.
  stereotactic radiosurgery : Pre-operative single fraction SRS
Period: Overall Study
Arm/Group | Pre-Operative SRS
Started | 6
Completed | 5
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Pre-OP SRS: SRS pre-operatively with the planned target volume defined as the tumor plus a 3-mm margin.
  therapeutic conventional surgery : Surgery of a single brain metastasis.
  stereotactic radiosurgery : Pre-operative single fraction SRS
Arm/Group | Pre-OP SRS
Number analyzed (Participants) | 6
Age Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Local Recurrence at the Surgical Site Within 12 Months After Stereotactic Radiosurgery (SRS)
Description: Number of patients with local recurrence at the surgical site within 12 months after stereotactic radiosurgery (SRS) as measured by magnetic resonance imaging (MRI). To determine local recurrence, we evaluated follow-up MRI's for reappearance of a lesion in exactly the same site in the brain as the first lesion(s).
Time Frame: Within 12 months after SRS
Population: Intent-to-treat; 1 patient was not included in this analysis as they were unable to undergo surgery after SRS.
Measure: Number; unit: Participants
Groups:
- Pre-Operative SRS: Stereotactic radiosurgery (SRS) will be administered pre-operatively as a single fraction with the planned target volume defined as the gross tumor volume plus a 3mm margin.
Arm/Group | Pre-Operative SRS
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Number of Patients Receiving Salvage Whole-brain Radiotherapy, Stereotactic Radiosurgery (SRS), or Surgery
Description: Number of patients receiving salvage whole-brain radiotherapy, stereotactic radiosurgery (SRS), or surgery
Time Frame: Within 24 months post-SRS
Population: Intent-to-treat; 1 patient was not included in this analysis as they were unable to undergo surgery after SRS.
Measure: Number; unit: participants
Arm/Group | Pre-Operative SRS
Number analyzed (Participants) | 5
participants | 2

3. Secondary Outcome: Volume of Adjacent Normal Brain Parenchyma Irradiated
Description: Volume of adjacent normal brain parenchyma irradiated during stereotactic radiosurgery (SRS).
Time Frame: At time of SRS
Population: Data for this outcome was not collected.
Arm/Group | Pre-Operative SRS
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Patients With New Brain Metastases Outside of the Pre-operative Stereotactic Radiosurgery (SRS) Site
Description: Number of patients with new brain metastases outside of the pre-operative stereotactic radiosurgery (SRS) site.
Time Frame: Within 24 months post-SRS
Population: Intent-to-treat; 1 patient was not included in this analysis as they were unable to undergo surgery after SRS.
Measure: Number; unit: participants
Arm/Group | Pre-Operative SRS
Number analyzed (Participants) | 5
participants | 2

5. Secondary Outcome: Quality of Life After Stereotactic Radiosurgery (SRS) as Measured by the Functional Assessment of Cancer Therapy-Brain (FACT-Br)
Description: Quality of life as measured by the change in FACT-Br scores from baseline. The FACT-Br (version 4) is comprised of the Functional Assessment of Cancer Therapy-General (FACT-G), a 27-item core questionnaire evaluating the domains of physical, family/social, emotional and functional well-being, with the addition of 23 brain cancer specific questions. The FACT-G total score is the sum of the four FACT-G domain scores. The Brain Cancer Subscale (BrCS) is the sum of 19 brain cancer specific questions. The FACT-Br Trial Outcome Index (TOI) is the sum of the BrCS score and the physical and family/social domain scores. The FACT-Br total score is the sum of the FACT-G total score and the BrCS score. Change score = score post-SRS minus the score at baseline. Positive change scores indicate improved quality of life.
Time Frame: Administered at baseline and every 3 months post-SRS
Population: Data for this outcome was erroneously not gathered.
Arm/Group | Pre-Operative SRS
Number analyzed (Participants) | 0

6. Secondary Outcome: Preservation of Neurocognitive Functioning as Measure by the Mini-Mental State Exam (MMSE)
Description: Cognition as measured by the change in the Mini-Mental State Exam (MMSE) scores from baseline. The MMSE is an 11-item measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall and language. The maximum score is 30. Change score = score post-SRS minus the score at baseline. Positive change scores indicate improved cognition.
Time Frame: Administered at baseline and every 3 months post-SRS
Population: Data for this outcome was erroneously not gathered.
Arm/Group | Pre-Operative SRS
Number analyzed (Participants) | 0

7. Secondary Outcome: Clinical Significance of Locally Recurrent Brain Metastases
Description: Number of patients with clinical significance (mass effect, cognitive functioning, and other symptoms) of locally recurrent brain metastases at the time of their occurrence.
Time Frame: 24 months post-SRS
Population: There are no patients for this analysis because none had a local recurrence.
Arm/Group | Pre-Operative SRS
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Patients Who Died Due to Neurological Causes
Description: Number of patients who died due to neurological causes defined as death attributable to the progression of neurological disease.
Time Frame: Within 24 months post-SRS
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Pre-Operative SRS
Number analyzed (Participants) | 6
participants | 0

9. Secondary Outcome: Overall Survival (OS)
Description: Time in months from the date of stereotactic radiosurgery (SRS) to the date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: 24 months after SRS
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pre-Operative SRS
Number analyzed (Participants) | 6
Months | 6.6 [3.5 to 13.2]

ADVERSE EVENTS:
Time Frame: 24 months
Description: The adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, and have been converted to CTCAE version 4.0 for entry into ClinicalTrials.gov.
Arm/Group | Pre-Operative SRS
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Operative SRS (N=6)
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes